CLINICAL TRIAL: NCT06390631
Title: Effect of CPAP on Respiratory Load and Lung Volume in Stable COPD
Brief Title: Effect of CPAP on Respiratory Load in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State Key Laboratory of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Yuan-Ming Luo, Professor, State Key Laboratory of Respiratory Disease
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020 No.38
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; CPAP; Diaphragm EMG
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: CPAP treatment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CPAP treatment (Experimental): CPAP treatment in COPD patients
  Interventions: Device: Continuous Positive Airway Pressure

INTERVENTIONS:
Device: Continuous Positive Airway Pressure — Patients with COPD were recruited to breath under the atmosphere pressure and different levels of CPAP (4, 6, 8 and 10 cm H2O).

SUMMARY:
Both intrinsic positive end expiratory pressure (PEEPi) and dynamic hyperinflation are considered as inspiratory loads which increase work of breathing in patients with COPD. The application of extrinsic positive end expiratory pressure (PEEPe) supplied by CPAP has been claimed to reduce inspiratory load based on change in esophageal pressure which could be significantly affected by change in lung volume and airflow. The investigator hypothesized that CPAP could increase respiratory load because it increases lung volume.

DETAILED DESCRIPTION:
Objective: To assess the effect of CPAP on respiratory load and lung volume in stable COPD. Methods: Patients with COPD were recruited to breath under the atmosphere pressure and different levels of CPAP (4, 6, 8 and 10 cm H2O). Diaphragm EMG, esophageal pressure (Pes) and transdiaphragmatic pressure (Pdi) were recorded using balloon esophageal electrode catheter (Yinghui, Guangzhou, China). End inspiratory lung volume (EILV) was measured directly from a pneumotachograph combined with a three way valve under the different CPAP levels. Sensation of breathing difficulty was also assessed. In an additional study, the effect of airflow on pressure was investigated by a physical mode.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate after informed consent
2. Males and females, any race and aged 40-80 years
3. GOLD II-IV COPD (post-bronchodilator FEV1 < 80 % of the predicted normal, and a post-bronchodilator FEV1/FVC < 0.70)

Exclusion Criteria:

1. Patients recovering from acute exacerbation less than 4 weeks.
2. Patients with concomitant pulmonary disease (e.g. lung fibrosis, interstitial lung disorder).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-09 (Actual)

PRIMARY OUTCOMES:
Diaphragm EMG | Around 5 minutes signals under the atmosphere pressure and different levels of CPAP (4, 6, 8 and 10 cm H2O) were recorded.
  assessment of the electrical activity of the diaphragm (EMG-di)
Lung volume | 1-3 minutes after each CPAP level (0, 4, 6, 8 and 10 cm H2O)
  measurement of end inspiratory lung volume (EILV)
Intrinsic positive end expiratory pressure (PEEPi) | Around 5 minutes signals under the atmosphere pressure and different levels of CPAP (4, 6, 8 and 10 cm H2O) were recorded.
  PEEPi was calculated from the negative deflection in Pes from the onset of inspiratory effort to the point of zero flow during spontaneous breathing.
Inspiratory pressure | Around 5 minutes signals under the atmosphere pressure and different levels of CPAP (4, 6, 8 and 10 cm H2O) were recorded.
  assessment of esophageal pressure and transdiaphragmatic pressure by caculating tidal variations in Pes (∆Pes) and Pdi (∆Pdi) relatived to initiation of effort.
Inspiratory work | Around 5 minutes signals under the atmosphere pressure and different levels of CPAP (4, 6, 8 and 10 cm H2O) were recorded.
  the pressure-time product of the respiratory muscles (PTPes/min) and of the diaphragm (PTPdi/min) were calculated under the Pes and Pdi versus time curve and expressed per minute.
Sensation of breathing effort | 5 minutes after each CPAP level (0, 4, 6, 8 and 10 cm H2O)
  Using questionnaire to assess the sensation of breathing effort. Sensation of breath effort of CPAP use was divided into three types corresponding to -1, 0, 1 score respectively, 0 refers to the same sensation as the feeling of breathing at the atmosphere without CPAP; 1 refers to the more difficult sensation to breath at the CPAP condition than at the atmosphere.; -1 refers to the easier sensation to breath at the CPAP condition than at the atmosphere.

SECONDARY OUTCOMES:
Respiratory rate (RR) | Around 5 minutes signals under the atmosphere pressure and different levels of CPAP (4, 6, 8 and 10 cm H2O) were recorded.
  assessment of respiratory rate (RR)
Tidal volume (Vt) | Around 5 minutes signals under the atmosphere pressure and different levels of CPAP (4, 6, 8 and 10 cm H2O) were recorded.
  assessment of tidal volume
Minute ventilation (VE) | Around 5 minutes signals under the atmosphere pressure and different levels of CPAP (4, 6, 8 and 10 cm H2O) were recorded.
  assessment of minute ventilation
Peak inspiratory flow rate | Around 5 minutes signals under the atmosphere pressure and different levels of CPAP (4, 6, 8 and 10 cm H2O) were recorded.
  assessment of peak inspiratory flow rate
Expiratory muscle EMG | Around 5 minutes signals under the atmosphere pressure and different levels of CPAP (4, 6, 8 and 10 cm H2O) were recorded.
  assessment of the electrical activity of the internal oblique muscle (EMG-obl) and the rectus muscle (EMG-rec)
Expiratory pressure | Around 5 minutes signals under the atmosphere pressure and different levels of CPAP (4, 6, 8 and 10 cm H2O) were recorded.
  The change in Pga resulting from the contraction of the abdominal muscles during expiration was analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Yuanming Luo, PHD, Principal Investigator — Guangzhou Medical University
Locations (1):
- Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared after the paper of this study publishing.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be shared after the paper of this study publishing.
Access Criteria: After the paper of this study publishing